CLINICAL TRIAL: NCT02581514
Title: Algorithm for the Early Diagnosis and Treatment of Patients With Eosinophilia
Brief Title: Eosinophilia Diagnosis
Acronym: EOSINOPHILIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I14028/EOSINOPHILIM
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Hypereosinophilic Syndrome
Keywords: decision algorithm
MeSH Terms: conditions — Hypereosinophilic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Algorithm (Experimental): Eosinophilia is assessed following the diagnosis algorithm
  Interventions: Other: Scheduled exams and diagnosis

INTERVENTIONS:
Other: Scheduled exams and diagnosis — Scheduled exams and diagnosis circuit as imposed by the algorithm

SUMMARY:
Eosinophilia, defined by a blood eosinophil granulocytes rate greater than 500 / mm3, is frequently encountered in internal medicine.

Its causes are varied: atopy, drug allergies, parasitic infections, autoimmune diseases and solid neoplasias. Over 200 etiologies have been reported, some difficult to diagnose and can be life-threatening Eosinophilia can be a diagnostic dilemma, as the etiologies are extensive and varied.

The aim of this study is to assess the feasibility of a diagnostic approach based on a decision algorithm in a group of patients with eosinophilia.

We assume that a procedure with a hierarchy of additional tests would increase the frequency of diagnosed cases while decreasing the time to diagnosis.

This procedure defined by an algorithm would even reduce the number of tests necessary to reach a diagnosis.

DETAILED DESCRIPTION:
Eosinophilia, defined by a blood eosinophil granulocytes rate greater than 500 / mm3, is frequently encountered in internal medicine.

Its causes are varied: atopy, drug allergies, parasitic infections, autoimmune diseases and solid neoplasias. Over 200 etiologies have been reported, some difficult to diagnose and can be life-threatening

Eosinophilia can be a diagnostic dilemma, as the etiologies are extensive and varied.

The aim of this study is to assess the feasibility of a diagnostic approach based on a decision algorithm in a group of patients with eosinophilia.

The contribution to the diagnosis of a hierarchical strategy for prescribing additional tests , based on clinical examination as well as some simple diagnostic tests, has never been evaluated

We assume that a procedure with a hierarchy of additional tests would increase the frequency of diagnosed cases while decreasing the time to diagnosis.

This procedure defined by an algorithm would even reduce the number of tests necessary to reach a diagnosis.

All types of patients are tacked into account: those coming from the university hospital, referred by general practitioners or by other hospitals.

In addition we address the internal medicine patients ,but also those of Hematology and Infectious Diseases. A comparison of these various groups would be relevant, since disorders that may be different.

Once enrolled, the patient is drived by the investigator through the various steps and exams imposed by the algorithm.

Indeed, during 5 months (Day1 5, 43, 71 , 85 , 99 ,113 and month 5), patient is asked to comply to the various exams and assessment imposed by the algorithm and that should lead to a diagnosis

ELIGIBILITY:
Inclusion Criteria:

1. Patient having one of the three following criteria:

   * hypereosinophilia> 1500 / mm3, checked on at least two samples (interval between 2 samples at the discretion of the clinician)
   * or hypereosinophilia> 500 cells / mm3 and organ damage with infiltration NCB proven by pathological examination,
   * or hypereosinophilia> 500 cells / mm3 and found consistently for at least six months (present on all controls carried out before inclusion).
2. Patient affiliated or beneficiary of a social security system
3. Patient who signed the informed consent

Exclusion Criteria:

1. Patient with solid tumors known (under chemotherapy or planned)
2. Patient unable to understand or to adhere to the Protocol
3. Patient unable to give consent
4. Pregnant or breastfeeding women
5. Patient already participating in an interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients having correctly follow the diagnosis algorithm | 5 months
  This outcome measure how many patients have correctly followed the diagnosis algorithm

SECONDARY OUTCOMES:
Rate of diagnosis | 5 months
  Evaluate the rate of diagnosis using our diagnosis algorithm
Assess the time to diagnosis | 5 months
  Assess the time to diagnosis
Description of diagnosis | 5 months
  To compare the diagnosis found in our study to the published cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Holy BEZANAHARY, Principal Investigator — University Hospital, Limoges
Locations (1):
- Médecine Interne A, Limoges, France